CLINICAL TRIAL: NCT04972721
Title: SELECT-LIFE (SELECT Follow-up Study to Evaluate Long-term Impact oF Anti-obEsity Medication)
Brief Title: SELECT-LIFE: A Research Study Looking at Long-term Effects of Semaglutide in People Who Took Part in the SELECT Cardiovascular Outcomes Trial
Acronym: SELECT-LIFE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: EX9536-4750; U1111-1255-5644 (Other: World Health Organization (WHO))
Record Dates: First submitted 2021-07-13; First posted 2021-07-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaire survey: Participants of the SELECT trial (EX9536-4388 ) are invited to transition to SELECT-LIFE (follow-up study) when SELECT ends.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — The study is non-interventional with no study-specific treatment during the study and the patients will be treated as per Treating Physician's and patient's own discretion.

SUMMARY:
Participants are being asked to participate in SELECT-LIFE study because participants take part in the SELECT trial.

SELECT-LIFE study is a survey-based study that will start when the SELECT trial ends.

SELECT-LIFE looks at the long-term effects of participants taking part in the SELECT trial including the trial medicine participants have been taking.

When the SELECT trial ends, participants will no longer get the medicine participants got in the study, even if participants decide to take part in the SELECT-LIFE study.

Participants will not get any specific treatment or medicine as part of the SELECT-LIFE study, and participants will be treated as participants normally would by their own doctor.

The SELECT-LIFE study will last for up to 10 years after SELECT trial ends, and participants will be asked to fill in a questionnaire about their health every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Randomized into the SELECT clinical trial (EX9536-4388) and has not withdrawn consent, regardless of level of participation, dose achieved or treatment discontinuation.
* Signed SELECT-LIFE consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).

Exclusion criteria:

* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of the SELECT trial (EX9536-4388 ) are invited to transition to SELECT-LIFE (follow-up study) when SELECT ends.
Sampling Method: Non-Probability Sample
Enrollment: 3439 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2025-08-25 (Actual)

PRIMARY OUTCOMES:
Time to all-cause death | From P-FUa (is the end of trial visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to 120 months)
  Measured in months
Time to first occurrence of a composite consisting of: All-cause death, non-fatal myocardial infarction and non-fatal stroke | From P-FUa (is the end of trial visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to 120 months)
  Measured in months
Time to first occurrence of non-fatal myocardial infarction | From P-FUa (is the end of trial visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to 120 months)
  Measured in months
Time to first occurrence of non-fatal stroke | From P-FUa (is the end of trial visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to 120 months)
  Measured in months
Time to diagnosis of type 2 diabetes | From P-FUa (is the end of trial visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to 120 months)
  Measured in months
Time to first occurrence of any type of cancer | From P-FUa (is the end of trial visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to 120 months)
  Measured in months
Time to first occurrence of a composite of obesity related cancer defined by WHO | From P-FUa (is the end of trial visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to 120 months)
  Measured in months
Time to first occurrence of knee replacement | From P-FUa (is the end of trial visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to 120 months)
  Measured in months
Time to first occurrence of bariatric surgery | From P-FUa (is the end of trial visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to 120 months)
  Measured in months
Time to first occurrence of anti-obesity medical treatment | From P-FUa (is the end of trial visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to 120 months)
  Measured in months
Time to first occurrence of use of continuous positive airways pressure (CPAP) device | From P-FUa (is the end of trial visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to 120 months)
  Measured in months
Total number of myocardial infarctions | From P-FUa (is the end of trial visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to 120 months)
  Measured in months
Total number of strokes | From P-FUa (is the end of trial visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to 120 months)
  Measured in months
Change in body weight from V-EOT (is the end of treatment visit in SELECT) to biannual assessments, (year 1-10) | From V-EOT (is the end of treatment visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to120 months)
  Measured in Kg
Change in Patient reported quality of life questionnaire (EQ-5D-5L) from V-EOT (is the end of treatment visit in SELECT) to biannual assessments, (year 1-10) | From V-EOT (is the end of treatment visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to120 months)
  EQ-5D-5L score The EQ-5D-5L questionnaire will be used to estimate the impact on subjects' health-related quality of life and provides a description of subjects' problems by dimensions (descriptive system), a score for overall self-rated health (visual analogue scale [VAS]) as well as an index score (EQ-5D-5L index). EQ-5D index score range: 0 to 1 and EQ-5D-VAS: range 0 to 100. A higher score indicates better self reported health status.
Total Days of hospitalisation from P-FU (is the end of trial visit in SELECT) to biannual assessments, (year 1-10) | From P-FU(is the end of trial visit in SELECT) (Day 1) to End of Study in SELECT-LIFE (up to120 months)
  Days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (38):
- Master Centre for USA, Plainsboro, New Jersey, United States
- Master Centre for Algeria, Algiers, Algeria
- Master Centre for Argentina, Prov. de Buenos Aires, Argentina
- Master Centre for Australia, North Sydney, New South Wales, Australia
- Brazil (15):
  - Cárdio Pulmonar da Bahia, Salvador, Estado de Bahia
  - Hospital do Coração do Brasil, Brasília, Federal District
  - Eurolatino Medical Research Center, Uberlândia, Minas Gerais
  - Núcleo de Pesquisa Clínica S/S, Curitiba, Paraná
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - AngioCor Blumenau, Blumenau, Santa Catarina
  - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - CIP Centro Integrado de Pesquisas do Hospital de Base, São José do Rio Preto, São Paulo
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas, São Paulo, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo
  - Departamento de Gastroenterologia - HCFMUSP, São Paulo, São Paulo
  - Instituto do Coração - HCFMUSP, São Paulo, São Paulo
  - Master Centre for Brazil, Säo Paulo, São Paulo
  - Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
- Master Centre for Canada, Mississauga, Ontario, Canada
- Novo Nordisk Croatia Ltd., Zagreb, Croatia
- Master Centre for Denmark, Copenhagen S, Denmark
- Master Centre for Finland, Espoo, Finland
- Master Centre for Germany PMS, Mainz, Germany
- Master Centre for Greece, Vouliagment, Greece
- Master centre for India, Bangalore, India
- Master Centre for Ireland, Dublin, Ireland
- Master Centre for Italy, Rome, Italy
- Master Centre for Japan, Tokyo, Japan
- MAster Centre for Latvia, Marupes, Latvia
- Master Centre for Malaysia, Selangor Darul Ehsan, Malaysia
- Master Centre Netherlands, Alphen aan den Rijn, Netherlands
- Master Centre for Norway, Rud, Norway
- Master Centre for South Africa, Sandton, Gauteng, South Africa
- Master Centre for Sweden, Malmo, Sweden
- Master Centre for Tawain, Taipei, Taiwan
- Master Centre for Thailand, Bangkok, Thailand
- Master Centre for United Kingdom, Gatwick, West Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com